CLINICAL TRIAL: NCT01222533
Title: A Multicenter, Randomised, Placebo- and Active-controlled, 5 Way, Crossover Trial to Characterise the Pharmacokinetics and Evaluate the Bronchodilator Efficacy and Safety of Once-daily Tiotropium Delivered (Double-blind) From the Respimat Inhaler as Solution for Inhalation (1.25, 2.5, 5 mcg or Placebo) and as Inhalation Powder (18mcg) From the HandiHaler (Open Label) After 4 Week-treatment Periods in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium Respimat Pharmacokinetic Study in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.458; 2009-016251-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (5):
- Tiotropium low (Experimental): Tiotropium inhalation solution low dose
  Interventions: Drug: Tiotropium low
- Tiotropium medium (Experimental): Tiotropium inhalation solution medium dose
  Interventions: Drug: Tiotropium medium
- Tiotropium high (Experimental): Tiotropium inhalation solution high dose
  Interventions: Drug: Tiotropium high
- Tiotropium 18mcg (Active Comparator): Tiotropium inhalation powder 18mcg
  Interventions: Drug: Tiotropium 18mcg
- Tiotropium placebo (Placebo Comparator): Placebo inhalation solution
  Interventions: Drug: Tiotropium placebo

INTERVENTIONS:
Drug: Tiotropium medium — Tiotropium inhalation solution medium dose
  Arms: Tiotropium medium
Drug: Tiotropium low — Tiotropium inhalation solution low dose
  Arms: Tiotropium low
Drug: Tiotropium high — Tiotropium inhalation solution high dose
  Arms: Tiotropium high
Drug: Tiotropium 18mcg — Tiotropium inhalation powder 18mcg
  Arms: Tiotropium 18mcg
Drug: Tiotropium placebo — Placebo inhalation solution
  Arms: Tiotropium placebo

SUMMARY:
The purpose of this study is compare the effect of different doses of tiotropium delivered by the HandiHaler and Respimat device on lung function. Additionally, the study will investigate the pharmacokinetic profile of these different doses. Studying the pharmacokinetic profile shows what happens to the medication in the body over a period of hours and provides information on potential effects of the medication.

ELIGIBILITY:
Inclusion criteria:

1. All patient must sign an informed consent consistent with IInternational Conference on Harmonisation- Good Clinical Practice (ICH-GCP) guidelines and local legislation prior to any study-related procedures, including medication washout and restrictions.
2. Relatively stable, moderate to very severe Chronic Obstructive Pulmonary Disease (COPD)
3. Current or ex-smokers (smoking history of at least 10 pack years)
4. Able to perform lung function tests
5. Able to use study inhalers

Exclusion criteria:

1. Significant diseases other than COPD
2. Recent myocardial infarction, unstable or life-threatening cardiac arrhythmia, hospitalisation for cardiac failure.
3. Malignancy requiring resection, radiation therapy or chemotherapy within the last 5 years
4. History of asthma, life-threatening pulmonary obstruction, cystic fibrosis or clinically evident bronchiectasis 5 Active tuberculosis

6. History of alcohol or drug abuse 7. Pulmonary resection 8. Recent completion of a pulmonary rehabilitation program or current participation which will not be continued 9. Daytime oxygen therapy for more than 1 hour per day. 10. Use of other investigational drugs, restrictions on the use of some respiratory medications during the study period.

11. Current participation in another clinical trial 12. Pregnant or nursing women 13. Women of childbearing potential not using a highly effective method of contraception (e.g: implants, injectable, oral contraceptives)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- Belgium (3):
  - 205.458.32003 Boehringer Ingelheim Investigational Site, Genk
  - 205.458.32001 Boehringer Ingelheim Investigational Site, Ghent
  - 205.458.32002 Boehringer Ingelheim Investigational Site, Hasselt
- Denmark (3):
  - 205.458.45001 Boehringer Ingelheim Investigational Site, Copenhagen K
  - 205.458.45003 Boehringer Ingelheim Investigational Site, København NV
  - 205.458.45002 Boehringer Ingelheim Investigational Site, Odense C
- Finland (2):
  - 205.458.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.458.35802 Boehringer Ingelheim Investigational Site, Tampere
- 205.458.49001 Boehringer Ingelheim Investigational Site, Hanover, Germany
- Netherlands (2):
  - 205.458.31001 Atrium Medisch Centrum Parkstad, Heerlen
  - 205.458.31002 Ommelander ziekenhuis groep, locatie Lucas, Winschoten

REFERENCES:
- [Derived] Hohlfeld JM, Furtwaengler A, Konen-Bergmann M, Wallenstein G, Walter B, Bateman ED. Cardiac safety of tiotropium in patients with COPD: a combined analysis of Holter-ECG data from four randomised clinical trials. Int J Clin Pract. 2015 Jan;69(1):72-80. doi: 10.1111/ijcp.12596. Epub 2014 Dec 11. PMID 25496316
- [Derived] Hohlfeld JM, Sharma A, van Noord JA, Cornelissen PJ, Derom E, Towse L, Peterkin V, Disse B. Pharmacokinetics and pharmacodynamics of tiotropium solution and tiotropium powder in chronic obstructive pulmonary disease. J Clin Pharmacol. 2014 Apr;54(4):405-14. doi: 10.1002/jcph.215. Epub 2013 Nov 27. PMID 24165906

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Overall: Total number of patients randomised and treated in the study. This was a randomised 5-period crossover trial. 154 patients were randomised to one of 15 sequences and treated. The trial was blinded within the 4 Respimat treatments, but open for the HandiHaler treatment. Each of the 5 treatment regimens was taken for 4 weeks without washouts between treatment periods.
Period: Overall Study
Arm/Group | Study Overall
Started | 154 (Entered and treated.)
Received Placebo | 147
Received Tio R1.25 | 147
Received Tio R2.5 | 145
Received Tio R5 | 150
Received Tio HH18 | 146
Completed | 140 (Completed planned observation time (week 21))
Not Completed | 14
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 5
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: Total number of patients randomised and treated in the study.
Arm/Group | Study Overall
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 117

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration at Steady-state (Cmax,ss)
Description: Cmax,ss is the maximum measured concentration of tiotropium in plasma at steady-state.
Time Frame: Based on blood sampling for PK assessments done at 4 weeks at the following time points: 5 minutes (min) before study drug (baseline) and at 2 min , 5 min, 7 min, 9 min, 12 min, 15 min, 20 min, 30 min, 40 min, 1 hour (h), 2 h, 4 h and 6 h post dosing.
Population: Pharmacokinetic (PK) Set. This analysis set includes all patients in the treated set who had at least one blood sample drawn or one urine sample collected for PK analysis. Patients with an important protocol violation relevant to the PK population were excluded. No PK data for placebo. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Groups:
- Placebo: Matching Placebo once daily (qd) delivered by the Respimat inhaler
- Tio R1.25: Tiotropium inhalation solution 1.25 mcg delivered by the Respimat inhaler qd in the morning
- Tio R2.5: Tiotropium inhalation solution 2.5 mcg delivered by the Respimat inhaler qd in the morning
- Tio R5: Tiotropium inhalation solution 5 mcg delivered by the Respimat inhaler qd in the morning
- Tio HH18: Open-label tiotropium inhalation capsule 18 mcg delivered by the HandiHaler qd in the morning
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 104 | 110 | 113 | 113
pg/ml |  | 2.81 (53.0) | 5.07 (61.8) | 10.5 (66.4) | 12.9 (64.6)
Statistical Analysis 1: Comparison: Tio R5 vs Tio HH18; Test type: Non-Inferiority or Equivalence — The standard bioequivalence range of 80 to 125% was pre-specified for Cmax,ss in order to assess the relative systemic exposure following inhalation of Tio R5 compared to Tio HH18. Bioequivalence was not used as a surrogate for efficacy; p = 0.4423, ANOVA — Maximum of two one-sided p-values for geometric mean ratio being outside interval 80 percent to 125 percent; Geometric mean ratio (percentage) = 80.66, 90% CI [73.49 to 88.52], Standard Deviation 43.4 — Standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Area Under the Curve 0 to 6 Hours at Steady-state (AUC0-6h,ss)
Description: AUC0-6h,ss is the area under the concentration time curve of tiotropium in plasma over the time interval 0 to 6 hours post-dose at steady-state. AUC0-6h,ss was calculated using the linear up/log down algorithm.
Time Frame: as for outcome 1
Population: PK Set. No PK data for Placebo. The low number of non-missing AUC0-6h,ss results for the Tio R 1.25 and Tio R 2.5 cohorts is due to the exclusion of results below the limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/ml
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 22 | 76 | 107 | 113
pg*h/ml |  | 10.0 (25.3) | 12.8 (29.9) | 22.1 (47.8) | 28.4 (52.4)
Statistical Analysis 1: Comparison: Tio R5 vs Tio HH18; Test type: Non-Inferiority or Equivalence — The standard bioequivalence range of 80 to 125% was pre-specified for AUC0-6,ss in order to assess the relative systemic exposure following inhalation of Tio R5 compared to Tio HH18. Bioequivalence was not used as a surrogate for efficacy; p = 0.8683, ANOVA — Maximum of two one-sided p-values for geometric mean ratio being outside interval 80 percent to 125 percent; Geometric mean ratio (percentage) = 75.99, 90% CI [70.44 to 81.98], Standard Deviation 34.1 — Standard deviation is actually the geometric coefficient of variation

3. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) at the End of Each Treatment Period
Description: Defined as FEV1 measured just prior to the last administration of the morning dose of the randomised treatment. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: Full analysis set (FAS) with imputed data. FAS includes all patients in the treated set who have analysable data for at least one efficacy endpoint during the relevant crossover period.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 143 | 143 | 144 | 143 | 142
Liter | 1.345 (0.045) | 1.432 (0.045) | 1.446 (0.045) | 1.466 (0.045) | 1.473 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.087, 95% CI [0.060 to 0.114], Standard Error of Mean 0.014 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.101, 95% CI [0.074 to 0.128], Standard Error of Mean 0.014 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.121, 95% CI [0.094 to 0.148], Standard Error of Mean 0.014 — Tio R5-Placebo

4. Secondary Outcome: FEV1 Area Under the Curve 0 to 6 Hours (AUC0-6h) at the End of Each Treatment Period
Description: FEV1 AUC0-6h calculated from zero time to 6 hours using the trapezoidal rule divided by 6 hours. Trough FEV1 will be assigned to zero time. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: FAS with imputed data.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 143 | 143 | 144 | 143 | 142
Liter | 1.371 (0.046) | 1.535 (0.046) | 1.556 (0.046) | 1.562 (0.046) | 1.567 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.165, 95% CI [0.141 to 0.189], Standard Error of Mean 0.012 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.185, 95% CI [0.161 to 0.209], Standard Error of Mean 0.012 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.191, 95% CI [0.167 to 0.216], Standard Error of Mean 0.012 — Tio R5-Placebo

5. Secondary Outcome: FEV1 Area Under the Curve 0 to 3 Hours (AUC0-3h) at the End of Each Treatment Period
Description: FEV1 AUC0-3h calculated from zero time to 3 hours using the trapezoidal rule divided by 3 hours. Trough FEV1 will be assigned to zero time. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: FAS with imputed data.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 143 | 143 | 144 | 143 | 142
Liter | 1.366 (0.046) | 1.521 (0.046) | 1.546 (0.046) | 1.553 (0.046) | 1.558 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.155, 95% CI [0.130 to 0.180], Standard Error of Mean 0.013 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.180, 95% CI [0.155 to 0.205], Standard Error of Mean 0.013 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.187, 95% CI [0.162 to 0.211], Standard Error of Mean 0.013 — Tio R5-Placebo

6. Secondary Outcome: Trough Forced Vital Capacity (FVC) at the End of Each Treatment Period
Description: Defined as the pre-dose FVC measured just prior to the last administration of the morning dose of the randomised treatment. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: FAS with imputed data. One patient with missing FVC data in Placebo and Tio R2.5 period.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 142 | 143 | 143 | 143 | 142
Liter | 3.116 (0.077) | 3.254 (0.077) | 3.304 (0.077) | 3.352 (0.077) | 3.351 (0.077)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.138, 95% CI [0.083 to 0.194], Standard Error of Mean 0.028 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.188, 95% CI [0.133 to 0.244], Standard Error of Mean 0.028 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.236, 95% CI [0.180 to 0.292], Standard Error of Mean 0.028 — Tio R5-Placebo

7. Secondary Outcome: FVC AUC0-6h at the End of Each Treatment Period
Description: FVC AUC0-6h calculated from zero time to 6 hours using the trapezoidal rule divided by 6 hours. Trough FVC will be assigned to zero time. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: FAS with imputed data. One patient with missing FVC data in Placebo and Tio R2.5 period.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 142 | 143 | 143 | 143 | 142
Liter | 3.153 (0.079) | 3.436 (0.078) | 3.472 (0.078) | 3.488 (0.078) | 3.483 (0.079)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.283, 95% CI [0.241 to 0.326], Standard Error of Mean 0.022 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.319, 95% CI [0.276 to 0.362], Standard Error of Mean 0.022 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.335, 95% CI [0.292 to 0.378], Standard Error of Mean 0.022 — Tio R5-Placebo

8. Secondary Outcome: FVC AUC0-3h at the End of Each Treatment Period
Description: FVC AUC0-3h calculated from zero time to 3 hours using the trapezoidal rule divided by 3 hours. Trough FVC will be assigned to zero time. Means are adjusted for sequence, patients within sequences, period and treatment.
Time Frame: 4 weeks
Population: FAS with imputed data. One patient with missing FVC data in Placebo and Tio R2.5 period.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 142 | 143 | 143 | 143 | 142
Liter | 3.140 (0.078) | 3.421 (0.078) | 3.465 (0.078) | 3.479 (0.078) | 3.480 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25; Test type: Superiority or Other; Mean Difference (Final Values) = 0.281, 95% CI [0.236 to 0.325], Standard Error of Mean 0.023 — Tio R1.25-Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.324, 95% CI [0.279 to 0.369], Standard Error of Mean 0.023 — Tio R2.5-Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for sequence, patients within sequences, period and treatment; Mean Difference (Final Values) = 0.339, 95% CI [0.294 to 0.384], Standard Error of Mean 0.023 — Tio R5-Placebo

9. Secondary Outcome: FEV1 at Each Planned Time at the End of Each Treatment Period
Description: Means are adjusted for period, planned time, period*planned time, patient*planned time and patient*treatment*planned time.
Time Frame: 4 weeks
Population: FAS with imputed data.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 143 | 143 | 144 | 143 | 142
Liter
  Timepoint 0:00 (trough) | 1.349 (0.045) | 1.436 (0.045) | 1.450 (0.045) | 1.470 (0.045) | 1.477 (0.045)
  Timepoint 0:30 | 1.366 (0.046) | 1.501 (0.046) | 1.522 (0.046) | 1.541 (0.046) | 1.554 (0.046)
  Timepoint 1:00 | 1.371 (0.046) | 1.529 (0.046) | 1.552 (0.046) | 1.560 (0.046) | 1.571 (0.046)
  Timepoint 2:00 | 1.375 (0.046) | 1.543 (0.046) | 1.573 (0.046) | 1.572 (0.046) | 1.571 (0.046)
  Timepoint 3:00 | 1.375 (0.047) | 1.556 (0.047) | 1.582 (0.047) | 1.584 (0.047) | 1.580 (0.047)
  Timepoint 4:00 | 1.374 (0.047) | 1.557 (0.047) | 1.575 (0.047) | 1.578 (0.047) | 1.582 (0.047)
  Timepoint 5:00 | 1.394 (0.047) | 1.562 (0.047) | 1.571 (0.047) | 1.579 (0.047) | 1.588 (0.047)
  Timepoint 6:00 | 1.375 (0.047) | 1.536 (0.048) | 1.551 (0.047) | 1.558 (0.047) | 1.570 (0.048)

10. Secondary Outcome: FVC at Each Planned Time at the End of Each Treatment Period
Description: as for outcome 9
Time Frame: 4 weeks
Population: FAS with imputed data. One patient with missing FVC data in Placebo and Tio R2.5 period.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 142 | 143 | 143 | 143 | 142
Liter
  Timepoint 0:00 (trough) | 3.118 (0.076) | 3.255 (0.076) | 3.307 (0.076) | 3.356 (0.076) | 3.351 (0.076)
  Timepoint 0:30 | 3.131 (0.077) | 3.390 (0.077) | 3.435 (0.077) | 3.473 (0.077) | 3.496 (0.077)
  Timepoint 1:00 | 3.152 (0.078) | 3.449 (0.078) | 3.484 (0.078) | 3.488 (0.078) | 3.499 (0.078)
  Timepoint 2:00 | 3.146 (0.078) | 3.443 (0.078) | 3.489 (0.078) | 3.499 (0.078) | 3.487 (0.078)
  Timepoint 3:00 | 3.156 (0.078) | 3.466 (0.078) | 3.513 (0.078) | 3.516 (0.078) | 3.497 (0.078)
  Timepoint 4:00 | 3.161 (0.079) | 3.468 (0.079) | 3.495 (0.079) | 3.505 (0.079) | 3.501 (0.079)
  Timepoint 5:00 | 3.191 (0.079) | 3.459 (0.079) | 3.467 (0.079) | 3.501 (0.079) | 3.488 (0.079)
  Timepoint 6:00 | 3.168 (0.079) | 3.417 (0.079) | 3.470 (0.079) | 3.473 (0.079) | 3.469 (0.079)

11. Secondary Outcome: Area Under the Curve 0 to 1 Hour at Steady-state (AUC0-1h,ss)
Description: AUC0-1h,ss is the area under the concentration time curve of tiotropium in plasma over the time interval 0 to 1 hour post-dose at steady-state. AUC0-1h,ss was calculated using the linear up/log down algorithm.
Time Frame: as for outcome 1
Population: PK Set. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 61 | 97 | 112 | 113
pg*h/mL |  | 2.08 (32.3) | 3.16 (44.4) | 6.13 (58.3) | 7.79 (54.9)

12. Secondary Outcome: Time to Maximum Plasma Concentration at Steady-state (Tmax,ss)
Description: Tmax,ss is the time from dosing to the maximum concentration of tiotropium in plasma-venous blood at steady-state.
Time Frame: Based on blood sampling for PK assessments done at 4 weeks at the following time points: 5 min before first dosing of study drug (baseline) and at 2 min , 5 min, 7 min, 9 min, 12 min, 15 min, 20 min, 30 min, 40 min, 1 h, 2 h, 4 h and 6 h post dosing.
Population: PK Set. All patients with analysable data.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 104 | 110 | 113 | 113
hours |  | 0.100 [0.0330 to 2.00] | 0.0830 [0.0330 to 6.00] | 0.117 [0.0330 to 0.333] | 0.117 [0.0330 to 1.00]

13. Secondary Outcome: Amount of Drug Eliminated in Urine at Steady-state (Ae0-6h,ss)
Description: Total quantity of the analyte that is excreted in urine over the time interval 0 to 6 hours at steady state.
Time Frame: Based on urine sampling for PK assessments done at 4 weeks in the following intervals: -1 to 0 hour (h), 0 to 2 h and 2 to 6 h post-dosing.
Population: PK Set. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 108 | 110 | 107 | 109
ng |  | 88.7 (68.0) | 177 (68.0) | 387 (65.9) | 522 (53.8)

14. Secondary Outcome: Pre-dose Plasma Concentration at Steady-state (Cpre,ss)
Description: Cpre,ss is the measured concentration of tiotropium in plasma before dosing at steady-state.
Time Frame: Based on blood sampling for PK assessments done at 4 weeks at the following time point: 5 minutes (min) before first dosing of study drug (baseline)
Population: PK Set. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 5 | 19 | 74 | 85
pg/mL |  | 1.57 (43.1) | 1.39 (22.8) | 1.60 (35.8) | 1.71 (42.5)

15. Secondary Outcome: Renal Clearance at Steady-state (CL R,0-6h,ss)
Description: Renal clearance of the drug over the time interval 0 to 6 hours at steady-state. CL R,0-6h,ss was calculated as the quotient of Ae0-6h,ss and AUC0-6h,ss.
Time Frame: Based on blood and urine sampling for PK assessments done at 4 weeks over 6 h post dosing.
Population: PK Set. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 22 | 75 | 102 | 109
mL/min |  | 256 (32.1) | 277 (55.8) | 307 (39.6) | 310 (40.4)

16. Secondary Outcome: Minimum Plasma Concentration at Steady-state (Cmin,ss)
Description: Cmin,ss is the minimum measured concentration of tiotropium in plasma at steady-state.
Time Frame: as for outcome 12
Population: PK Set. All patients with analysable data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 0 | 103 | 110 | 113 | 113
pg/mL |  | 1.16 (14.5) | 1.25 (17.7) | 1.57 (32.3) | 1.76 (42.3)

17. Other Pre Specified Outcome: Maximum Heart Rate (HR)
Description: Maximum HR evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: ECGFAS - including all patients in the treated set for whom continuous 12 lead ECGs (Holter monitoring) were recorded on at least one occasion (pacemaker patients were excluded).
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
bpm
  Day 29 6.5 h(N=115,115,115,116,113) | 109.29 (15.23) | 109.57 (15.29) | 109.93 (15.47) | 109.34 (14.36) | 108.68 (14.28)
  Day 29 1st h(N=114,113,115,115,111) | 97.83 (13.65) | 99.20 (14.65) | 98.43 (14.68) | 97.16 (13.97) | 97.33 (13.00)
  Day 26 6.5 h(N=115,110,113,110,112) | 108.35 (16.32) | 107.37 (14.04) | 108.90 (15.85) | 107.65 (16.37) | 109.57 (14.70)
  Day 26 1st h(N=115,109,113,107,109) | 91.73 (12.44) | 91.51 (12.87) | 92.59 (15.40) | 91.60 (12.07) | 92.74 (12.75)

18. Other Pre Specified Outcome: Mean Heart Rate (HR)
Description: Mean HR evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
bpm
  Day 29 6.5 h(N=115,115,115,116,113) | 76.97 (10.39) | 76.37 (10.69) | 77.75 (10.95) | 76.87 (10.82) | 77.31 (10.45)
  Day 29 1st h(N=114,113,115,115,111) | 73.87 (10.07) | 73.76 (10.60) | 74.39 (10.82) | 73.82 (11.06) | 73.71 (9.80)
  Day 26 6.5 h(N=115,110,113,110,112) | 75.76 (10.88) | 75.00 (10.87) | 76.25 (12.00) | 75.35 (10.86) | 75.81 (10.39)
  Day 26 1st h(N=115,109,113,107,109) | 70.75 (10.20) | 70.33 (10.66) | 71.11 (11.93) | 70.67 (10.77) | 70.21 (9.58)

19. Other Pre Specified Outcome: SVPB Total
Description: The outcome measure describes the number of patients with a Supraventricular Premature Beat (SVPB) event evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 109 | 112 | 109 | 108 | 107
  Day 29 1st h | 83 | 79 | 75 | 84 | 75
  Day 26 6.5 h | 111 | 103 | 106 | 98 | 105
  Day 26 1st h | 82 | 74 | 75 | 62 | 66

20. Other Pre Specified Outcome: SVPB Runs
Description: The outcome measure describes the number of patients with a Supraventricular Premature Beat (SVPB) run evaluated over the entire 6.5 h Holter monitoring period. Runs were defined as at least 3 premature beats in a row. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 47 | 36 | 44 | 34 | 39
  Day 29 1st h | 9 | 16 | 8 | 5 | 6
  Day 26 6.5 h | 35 | 34 | 29 | 36 | 34
  Day 26 1st h | 12 | 6 | 9 | 11 | 10

21. Other Pre Specified Outcome: SVPB Pairs
Description: The outcome measure describes the number of patients with a Supraventricular Premature Beat (SVPB) pair evaluated over the entire 6.5 h Holter monitoring period. Pairs were defined as 2 consecutive premature beats in a row. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 48 | 52 | 55 | 49 | 53
  Day 29 1st h | 17 | 20 | 19 | 20 | 16
  Day 26 6.5 h | 41 | 46 | 29 | 42 | 45
  Day 26 1st h | 18 | 13 | 10 | 14 | 13

22. Other Pre Specified Outcome: SVPB Singles
Description: The outcome measure describes the number of patients with a Supraventricular Premature Beat (SVPB) single evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 109 | 112 | 109 | 108 | 107
  Day 29 1st h | 82 | 77 | 72 | 82 | 73
  Day 26 6.5 h | 111 | 102 | 106 | 98 | 105
  Day 26 1st h | 78 | 74 | 74 | 61 | 64

23. Other Pre Specified Outcome: VPB Total
Description: The outcome measure describes the number of patients with a Ventricular Premature Beat (VPB) event evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 91 | 99 | 90 | 96 | 96
  Day 29 1st h | 59 | 63 | 58 | 50 | 59
  Day 26 6.5 h | 92 | 82 | 83 | 89 | 88
  Day 26 1st h | 59 | 49 | 49 | 49 | 56

24. Other Pre Specified Outcome: VPB Runs
Description: The outcome measure describes the number of patients with a Ventricular Premature Beat (VPB) run evaluated over the entire 6.5 h Holter monitoring period. Runs were defined as at least 3 premature beats in a row. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 3 | 5 | 4 | 10 | 9
  Day 29 1st h | 0 | 3 | 2 | 2 | 1
  Day 26 6.5 h | 8 | 7 | 8 | 9 | 9
  Day 26 1st h | 0 | 2 | 1 | 4 | 3

25. Other Pre Specified Outcome: VPB Pairs
Description: The outcome measure describes the number of patients with a Ventricular Premature Beat (VPB) pair evaluated over the entire 6.5 h Holter monitoring period. Pairs were defined as 2 consecutive premature beats in a row. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 24 | 19 | 21 | 16 | 22
  Day 29 1st h | 8 | 6 | 6 | 6 | 7
  Day 26 6.5 h | 24 | 20 | 19 | 21 | 22
  Day 26 1st h | 7 | 10 | 7 | 6 | 10

26. Other Pre Specified Outcome: VPB Singles
Description: The outcome measure describes the number of patients with a Ventricular Premature Beat (VPB) single evaluated over the entire 6.5 h Holter monitoring period. The arrhythmia variables were pre-specified for day 29 and analysed post-hoc for day 26. The lines "Day 29 1st h" and "Day 26 1st h" are related to the interval 0 h to 1 h, i.e. the first hour after dosing.
Time Frame: 6.5 hours (including pre dose)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Number analyzed (Participants) | 115 | 115 | 115 | 116 | 113
participants
  Day 29 6.5 h | 91 | 99 | 89 | 94 | 96
  Day 29 1st h | 59 | 63 | 58 | 50 | 58
  Day 26 6.5 h | 92 | 82 | 81 | 88 | 88
  Day 26 1st h | 59 | 49 | 48 | 49 | 55

ADVERSE EVENTS:
Time Frame: 4 weeks + 30 days if in last period
Arm/Group | Placebo | Tio R1.25 | Tio R2.5 | Tio R5 | Tio HH18
Serious Adverse Events (participants affected / at risk) | 3/147 | 2/147 | 0/145 | 3/150 | 2/146
Other Adverse Events (participants affected / at risk) | 20/147 | 11/147 | 4/145 | 16/150 | 10/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Tio R1.25 (N=147) | Tio R2.5 (N=145) | Tio R5 (N=150) | Tio HH18 (N=146)
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Tio R1.25 (N=147) | Tio R2.5 (N=145) | Tio R5 (N=150) | Tio HH18 (N=146)
Nasopharyngitis (Infections and infestations) | 6 | 9 | 2 | 14 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication